CLINICAL TRIAL: NCT03870581
Title: Artificial Intelligence-based Social Software Management Model to Improve Warfarin Anticoagulation Therapy: a Prospective, Single-blind, Randomized Control Trial
Brief Title: AI-based Social Software to Manage wARfarin Therapy
Acronym: AI-SMART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wuhan Asia Heart Hospital (Other)
Responsible Party: Principal Investigator, Litao Zhang, MD, Head of anticoagulation clinic, Wuhan Asia Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-P-012
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Anticoagulant-induced Bleeding; Warfarin Sodium Causing Adverse Effects in Therapeutic Use
Keywords: Artificial intelligence; social software; warfarin; anticoagulation therapy; INR

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants did not know whether they were assigned to AI-SMART group or Human-SMART group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-SMART group (Experimental): Participants' warfarin therapy were guided by an AI-based miniprogram embedded in the Wechat social software.
  Interventions: Behavioral: AI-based social software management model
- Human-SMART group (Active Comparator): Participants' warfarin therapy were guided by an human-based miniprogram embedded in the Wechat social software.
  Interventions: Behavioral: Human-based social software management model

INTERVENTIONS:
Behavioral: AI-based social software management model — a AI-based miniprogram, embedded in the Wechat social software, to manage participants' warfarin therapy, such as dose adjustment, INR monitoring alert, etc.
  Other Names: Warfarin Helper-AI
  Arms: AI-SMART group
Behavioral: Human-based social software management model — a Human-based miniprogram, embedded in the Wechat social software, to manage participants' warfarin therapy, such as dose adjustment, INR monitoring alert, etc.
  Other Names: Warfarin Helper
  Arms: Human-SMART group

SUMMARY:
The investigators have demonstrated that social software could improve warfarin therapy quality by Human management. however,the efficiency of management will decline if patients' number expands huge. So it is needed that a human-like and automatic management tool could replace the human work. The aim of this study is to evaluate whether an AI-based social software management model could replace human to guide warfarin therapy.

DETAILED DESCRIPTION:
1. The investigators have developed an AI-based miniprogram, and embedded in the Wechat social application.
2. The investigators invited patients receiving warfarin therapy to participant this randomized controlled trial .
3. Participants were randomized to the experimental group and control group in a ratio of 1:1.
4. Participants' warfarin therapy were managed by an AI-based social miniprogram and a Human-based social miniprogram respectively.
5. International normalized ratio(INR) was monitored once a month at least, and the time in therapeutic range was calculated to evaluate the warfarin anticoagulation quality.
6. Participants were followed-up for 24 months, and clinical events, including major bleedings and thrombotic events were recorded during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Atrial fibrillation
* Patients with Mechanical valve replacement
* Patients receiving warfarin therapy

Exclusion Criteria:

* Plan to stop warfarin therapy within 1 years
* Bleeding within 3 months
* Refuse to participate in this study
* Other conditions that the physician considers inappropriate for participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Time in therapeutic range | 24 months
  Calculated Time of international normalized ratio in therapeutic range
INR variability | 24 months
  coefficient of variation of international normalized ratio (INR)

SECONDARY OUTCOMES:
Bleeding events | 24 months
  Including Cerebral hemorrhage, gastrointestinal bleeding and other major bleeding
Thrombotic events | 24 months
  Including stroke, deep vein thrombosis,Pulmonary embolism,Peripheral arterial embolism, et.al

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - WAHH, Wuhan, Hubei
  - Wuhan Asia Heart Hospital, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR